CLINICAL TRIAL: NCT07217522
Title: Rutgers University Study of the Genetics of Pulmonary Hypertension
Acronym: RUGCC-PH
Status: Recruiting | Type: Observational
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Tara Matise, Ph.D., Distinguished Professor, Rutgers, The State University of New Jersey
Other Study IDs: Pro2025001041
Record Dates: First submitted 2025-10-14; First posted 2025-10-16 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Pulmonary Hypertension; Pulmonary Arterial Hypertension; Pulmonary Arterial Hypertension (PAH) (WHO Group 1 PH); Pulmonary Arterial Hypertension Associated With Connective Tissue Disease; Pulmonary Arterial Hypertension Associated With Connective Tissue Disease (Disorder); Pulmonary Arterial Hypertension Associated With Schistosomiasis (Disorder); Pulmonary Arterial Hypertension of Congenital Heart Disease; Pulmonary Arterial and Chronic Thromboembolic Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension | interventions — Health Surveys

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pulmonary hypertension cases: Study participants who have been diagnosed with any form of pulmonary hypertension, either currently or in the past.
  Interventions: Genetic: Saliva sample; Other: Health surveys
- Pulmonary hypertension controls: Study participants who have not been diagnosed with any form of pulmonary hypertension, either currently or in the past.
  Interventions: Genetic: Saliva sample; Other: Health surveys

INTERVENTIONS:
Genetic: Saliva sample — Saliva sample is sent via prepaid US Mail for DNA extraction
Other: Health surveys — Health surveys are filled out online in the study portal.

SUMMARY:
The goal of this observational study is to learn more about how genes impact the risk of pulmonary hypertension. Anyone 18 or older living in the US is eligible, and a diagnosis of PH is NOT required. Study participation is online, and it takes about 20 minutes to complete health surveys and request a saliva collection kit sent through US mail. In return, study participants may opt to receive information about their genetic ancestry at no cost.

DETAILED DESCRIPTION:
This is an online research study to learn more about how genes affect the risk of pulmonary hypertension. No office visit is required and in return, participants may receive information about their genetic ancestry for free. Population-based echocardiography surveys show that pulmonary hypertension (PH) affects roughly 2-3 % of community-dwelling adults and becomes more common with age. This study will increase our understanding of the genetic basis of breast cancer, which is a crucial step in drug development to improve current treatment options. The study investigators seek a diverse population because diversity among participants maximizes the usefulness of the data. Participants will use our online study portal to answer questions about their health and provide their DNA via a saliva sample using a pre-paid mailer. Participation takes approximately 20 minutes. Participants will be invited to share data from their electronic health records, but this is not required for study participation. The study investigators keep participants engaged with short monthly newsletters.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* currently living in the United States
* able to understand and follow written instructions in English
* have access to the internet and a computer, laptop, tablet or smart phone
* willing to provide written informed consent for participation
* willing to provide DNA via a saliva sample using a collection kit mailed to the study participant's home
* willing to complete a survey with questions about health related to the study of pulmonary hypertension.

Exclusion Criteria:

* Age 17 or below
* Not currently living in the United States
* Not able to participate in an online research study in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of anyone at least 18 years old who lives in the United States, including both individuals who have or had pulmonary hypertension and those who have not. Participants include males, females, non-binary, and all race-ethnic groups.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2025-08-23 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Genetic risk variants associated with pulmonary hypertension | 2 years
  Genetic factors will be measured through whole exome sequencing along with genotyping of common variants, and then correlated with pulmonary hypertension and pulmonary hypertension subtype.

CONTACTS AND LOCATIONS:
Overall Officials: Tara Matise, Ph.D., Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- Rutgers University, Piscataway, New Jersey 08854, Piscataway, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Informational website about the study — https://rugcc.rutgers.edu/pulmonary-hypertension/